CLINICAL TRIAL: NCT03934268
Title: A Cohort Study on the Prognosis of Neonatal KCNQ2 Gene-associated Epileptic Encephalopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: CHFudanU_NNICU12
Record Dates: First submitted 2019-04-29; First posted 2019-05-01 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Seizures; Seizure Disorder; Seizure Newborn; Seizures, Generalized; Epileptic Encephalopathy; Epileptic Encephalopathy, Neonatal-onset; Epileptic Encephalopathy, Infant-onset; KCNQ2
MeSH Terms: conditions — Seizures; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The researchers retained the neonates' or infants' 2ml serum as a biological sample for the Whole Exon Sequencing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- infants with seizure with KCNQ2 gene mutation.: Infants who met the inclusion criteria were enrolled in this study. The infants will get their own DNA sequencing results by WES technology. The researchers found that some of them carried mutations in the KCNQ2 gene. so they wanted to compare whether there were differences with or without KCNQ2 gene mutations in the efficacy of anticonvulsants or long-term neurodevelopment in different exposure groups.
  Interventions: Genetic: KCNQ2

INTERVENTIONS:
Genetic: KCNQ2 — The researchers extracted DNA from the baby's serum and sent it to WES to get the baby's total exon sequence.

SUMMARY:
The researchers hope to explore the etiological distribution and influencing factors of KCNQ2-related neonatal convulsions or refractory epileptic encephalopathy, and to improve the level of assessment, identification, intervention and shunt of KCNQ2-related convulsions. To formulate countermeasures and measures for prevention, management and health education.

DETAILED DESCRIPTION:
Convulsion is the most common clinical manifestation of neonatal central nervous system dysfunction. the incidence of convulsion is very high in neonatal period, especially in the first week after birth. the incidence of convulsion decreases gradually with the increase of age. The incidence of convulsion reported by Bassan et al was 1.5 ‰ ~ 3.5 ‰ in term infants and 10% ≤ 130% in premature infants. Most of the neonatal convulsions suggest that there are serious primary diseases in the body. in addition to hypoxic-ischemic encephalopathy, intracranial hemorrhage and infection, a large number of studies have proved that genetic factors play a key role in the occurrence of neonatal convulsions and epileptic encephalopathy in infants. Nearly 20% to 50% of neonatal convulsions are idiopathic convulsions. it has been thought that KCNQ2 gene, a potassium channel subunit located in 20q11.3, and KCNQ3 gene, another potassium channel subunit located in 8q24, are mutated. Is the molecular basis for some benign familial neonatal convulsions, Usually the prognosis is good, but with the expansion of the study sample, investigators found that KCNQ2 may be associated with refractory epileptic encephalopathy, and there are few international reports in this regard. The study of KCNQ2 gene has led to a new understanding of the etiology of neonatal convulsion. The researchers hope to explore the etiological distribution and influencing factors of KCNQ2-related neonatal convulsions or refractory epileptic encephalopathy, and to improve the level of assessment, identification, intervention and shunt of KCNQ2-related convulsions. To formulate countermeasures and measures for prevention, management and health education.

ELIGIBILITY:
Inclusion Criteria:

* Primary or initial convulsion
* Postnatal age <28 days.
* Seizure in the neonatal period
* Informed consent of parents

Exclusion Criteria:

* Seizure caused by congenital cerebral hypoplasia or multiple structural malformations.
* Seizure caused by other system-related syndromes.
* Seizure caused by perinatal or postpartum factors such as HIE, infection, intracranial hemorrhage, etc.

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The subjects came from sub-central hospitals and the newborns were hospitalized in the neonatal department for primary seizure.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of seizure in children with KCNQ2 within 28 days of age | From birth to under 28 days of age
  The investigators used WES to screen for neonatal onset seizure and calculated the incidence of KCNQ2 gene mutations in these neonates.

SECONDARY OUTCOMES:
Recurrence rate of KNCQ2 gene-related convulsion in children under 1 year of age | From birth to under 1 year of age
  Some neonates with seizure associated with KCNQ2 gene mutation will develop epileptic encephalopathy or syndrome at a later stage.
  The researchers calculated the probability of recurrent seizures or progression in neonates with seizure associated with KCNQ2 gene mutations within the age of one year.
Efficacy of first-line anticonvulsants in children with KCNQ2 gene-related convulsions | From the beginning of drug intervention to 72 hours after taking the drug.
  Some non-benign KCNQ2 gene-related convulsions require anticonvulsant intervention, and investigators hope to observe and obtain the effective rate of first-line anticonvulsant intervention. To determine whether the convulsion stopped or the frequency of convulsion decreased within 72 hours after taking the drug. If convulsions stop or the frequency of seizures decreases, drug intervention is considered effective.
Proportion of infants classified as having "developmental delay" (MDI <70 on BSID-III or either Language or Cognitive Score <70 on the Bayley-III) | The infants will be evaluated by bayley Neurodevelopment scale at the age of about two years.
  The investigators plan to use the bayley Neurodevelopmental scale to assess the neurodevelopmental status of infants with KCNQ2 gene-associated epileptic encephalopathy within 2 years of age.

CONTACTS AND LOCATIONS:
Overall Officials: Wenhao Zhou, Prof., Study Chair — Children Hospital of Fudan University
Locations (1):
- Children Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuersten M, Tacke M, Gerstl L, Hoelz H, Stulpnagel CV, Borggraefe I. Antiepileptic therapy approaches in KCNQ2 related epilepsy: A systematic review. Eur J Med Genet. 2020 Jan;63(1):103628. doi: 10.1016/j.ejmg.2019.02.001. Epub 2019 Feb 14. PMID 30771507
- [Background] Cornet MC, Sands TT, Cilio MR. Neonatal epilepsies: Clinical management. Semin Fetal Neonatal Med. 2018 Jun;23(3):204-212. doi: 10.1016/j.siny.2018.01.004. Epub 2018 Jan 31. PMID 29426806
- [Background] Reif PS, Tsai MH, Helbig I, Rosenow F, Klein KM. Precision medicine in genetic epilepsies: break of dawn? Expert Rev Neurother. 2017 Apr;17(4):381-392. doi: 10.1080/14737175.2017.1253476. Epub 2016 Nov 10. PMID 27781560
- [Background] Hani AJ, Mikati HM, Mikati MA. Genetics of pediatric epilepsy. Pediatr Clin North Am. 2015 Jun;62(3):703-22. doi: 10.1016/j.pcl.2015.03.013. PMID 26022171
- [Result] Manville RW, Abbott GW. Ancient and modern anticonvulsants act synergistically in a KCNQ potassium channel binding pocket. Nat Commun. 2018 Sep 21;9(1):3845. doi: 10.1038/s41467-018-06339-2. PMID 30242262
- [Result] Manville RW, Papanikolaou M, Abbott GW. Direct neurotransmitter activation of voltage-gated potassium channels. Nat Commun. 2018 May 10;9(1):1847. doi: 10.1038/s41467-018-04266-w. PMID 29748663